CLINICAL TRIAL: NCT03472547
Title: A Randomized, Controlled Study to Evaluate the Sensitizing Potential of CCP-020 (Diacerein 1%) Topical Ointment in Healthy Subjects Using a Repeat Insult Patch Test Design
Brief Title: A Study of Sensitizing Potential of Diacerein 1% Ointment in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Castle Creek Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCP-020-103
Record Dates: First submitted 2018-01-30; First posted 2018-03-21 (Actual); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — diacerein; Ointments

STUDY DESIGN:
Intervention Model Description: All subjects were exposed to diacerein 1% ointment, vehicle ointment, and 0.9% saline (negative control) at 3 randomly assigned, adjacent skin sites on the infrascapular area of the back 3 times weekly for 3 weeks (9 applications) during the Induction Phase, and one time during the Challenge Phase (10 times in total).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single cohort (Healthy Volunteers) (Experimental): diacerein 1% ointment
  Interventions: Drug: diacerein 1% ointment

INTERVENTIONS:
Drug: diacerein 1% ointment — All subjects were exposed to diacerein 1% ointment, vehicle ointment, and 0.9% saline (negative control) at 3 randomly assigned, adjacent skin sites on the infrascapular area of the back 3 times weekly for 3 weeks (9 applications) during the Induction Phase, and one time during the Challenge Phase (10 times in total).
  Other Names: CCP-020

SUMMARY:
Single center, randomized, controlled, evaluator blinded, within-subject study to evaluate the sensitization potential of diacerein 1% ointment under occlusive conditions on normal skin of healthy volunteer subjects.

DETAILED DESCRIPTION:
The study was designed to assess the sensitization potential of diacerein 1% ointment in comparison to vehicle ointment and 0.9% saline (negative irritant control) under occlusive patch conditions, at 3 randomly assigned, adjacent skin sites, 3 times weekly for 3 weeks (9 applications) during the Induction Phase, and one time during the Challenge Phase (10 times in total) for determining sensitization potential.

ELIGIBILITY:
Key Inclusion Criteria:

* Is a healthy male or female (to be confirmed by medical history);
* Is 18 years of age or older;
* In the case of a female of childbearing potential, is using two acceptable forms of birth control;
* In the case of a female of childbearing potential, has a negative urine pregnancy test (UPT) on Day 1 prior to randomization and are willing to submit to a UPT at the end of study (EOS);
* Is free of any systemic or dermatological disorder, which, in the opinion of the Investigator, will interfere with the study results or increase the risk of AEs;
* Is of any Fitzpatrick Skin Type or race, providing the skin pigmentation will allow discernment of erythema

Key Exclusion Criteria:

* Has any visible skin disease at the application site which, in the opinion of the Investigator, will interfere with the evaluation of the test site reaction;
* Is using systemic/topical corticosteroids within 3 weeks prior to and/or during the study, or systemic/topical antihistamines 72 hours prior to and during the study;
* Is not willing to refrain from using systemic/topical anti-inflammatory analgesics such as aspirin (occasional use of acetaminophen will be permitted);
* Is using medication which, in the opinion of the Investigator, will interfere with the study results;
* Is unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions or similar products on the back during the study;
* Has psoriasis and/or active atopic dermatitis/eczema;
* Has a known sensitivity or allergy to constituents of the materials being evaluated; including diacerein, mineral oil, petrolatum, cetyl alcohol, D&C Yellow #10 and/or ethyl paraben;
* Has damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site;
* Has received treatment for any type of internal cancer within 5 years prior to study entry;
* Has any known sensitivity to adhesives; and/or
* Has received any investigational drug(s) within 4 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Spellman, MD, Study Chair — Castle Creek Pharmaceuticals, LLC
Locations (1):
- TKL Research, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: skin patch test sites
Groups:
- Single Cohort (Healthy Volunteers): All subjects were exposed to diacerein 1% ointment, vehicle ointment, and 0.9% saline (negative control) at 3 randomly assigned, adjacent skin sites on the infrascapular area of the back 3 times weekly for 3 weeks (9 applications) during the Induction Phase, and one time during the Challenge Phase (10 times in total).
Period: Overall Study
Arm/Group | Single Cohort (Healthy Volunteers)
Started | 234; 702 skin patch test sites
Completed | 204; 612 skin patch test sites
Not Completed | 30; 90 skin patch test sites
Not completed — Withdrawal by Subject | 30

BASELINE CHARACTERISTICS:
Arm/Group | Single Cohort (Healthy Volunteers)
Number analyzed (Participants) | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176
  Male | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 214
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 166
  White | 68
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Observed Sensitization
Description: The determination of dermal sensitization potential was based on the recurrence of a cutaneous response at re-challenge that was equivalent or more severe than the cumulative irritation score observed during the challenge period.
  Cumulative irritation score is a visual score rating the degree of erythema, edema, and other signs of cutaneous irritation: Minimum = 0; Maximum = 6; higher score is worse outcome.
Time Frame: 56 days
Population: The evaluation of sensitization was based on all subjects who completed the Challenge Phase of the study.
Measure: Number; unit: Participants with Observed Sensitization
Groups:
- Observed Sensitization: All subjects were exposed to diacerein 1% ointment, vehicle ointment, and 0.9% saline (negative control) at 3 randomly assigned, adjacent skin sites on the infrascapular area of the back 3 times weekly for 3 weeks (9 applications) during the Induction Phase, and one time during the Challenge Phase (10 times in total).
Arm/Group | Observed Sensitization
Number analyzed (Participants) | 204
Participants with Observed Sensitization
  Diacerein 1% ointment | 0
  vehicle ointment | 0
  0.9% saline (negative control) | 0

ADVERSE EVENTS:
Time Frame: 56 days
Description: Adverse events were not assessed at a patch site-specific level.
Arm/Group | Single Cohort (Healthy Volunteers)
All-Cause Mortality (participants affected / at risk) | 0/234
Serious Adverse Events (participants affected / at risk) | 0/234
Other Adverse Events (participants affected / at risk) | 0/234

LIMITATIONS AND CAVEATS:
There were no limitations or caveats in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT03472547/Prot_SAP_000.pdf